CLINICAL TRIAL: NCT04675645
Title: Adherence to Hydroxyurea and Health-related Quality of Life in Patients With Sickle Cell Disease: An Intervention Study Using a Smartphone App (HU-Go)
Brief Title: Adherence to HU and HRQOL in Patients With Sickle Cell Disease: An Intervention Study Using HU-Go App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Sherif Badawy, MD, Assistant Professor, Department of Pediatrics, Division of Hematology, Oncology and Stem Cell Transplant, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 2015-761
Record Dates: First submitted 2016-08-17; First posted 2020-12-19 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Sickle Cell Disease; Sickle B+ Thalassemia; Sickle Beta Zero Thalassemia; Sickle Cell Hemoglobin C
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HU-Go app intervention arm (Other): Participants will use HU-Go app intervention arm for a total of 12 weeks.
  Interventions: Other: HU-Go app

INTERVENTIONS:
Other: HU-Go app — A novel multifunctional mobile app (HU-Go) to improve adherence to hydroxyurea in patients with sickle cell disease

SUMMARY:
This project addresses three important research questions. First, adolescents and young adults (AYA) with sickle cell disease (SCD) and their parents/caregivers will be engaged to inform the (1) domains of health-related quality of life (HRQOL) most important to them, (2) frequency at which they are willing to complete them, and (3) other procedures related to the use, uptake and effect of the HU-Go app as a tool to improve hydroxyurea (HU) adherence. Second, this study seeks to utilize novel modern mobile technology using a multi-functional personalized platform to improve adherence to HU and measure HRQOL in youth with SCD, using NIH-endorsed PROMIS® measures, based on a conceptual model with predefined behavioral targets and mediators. Third, we plan to assess HRQOL changes and identify modifiable behavioral strategies that could serve as surrogates or predictors for HU adherence. This real-time feedback might empower self-directed changes in behavior that could improve adherence to HU.

DETAILED DESCRIPTION:
Aim 1: Identify the needs, desires, concerns, and expectations of AYA patients with SCD and their parents/caregivers that will guide implementation of a mHealth tool, HU-Go, designed to improve adherence to HU. We will conduct semi-structured interviews with patients and their parents/caregivers. Transcripts will be independently coded and thematic analysis will be conducted.

Hypothesis 1: AYA patients with SCD and their parents/caregivers will identify specific features, content, and usability requirements of HU-Go.

Aim 2: Assess the longitudinal relationship of HU adherence to HRQoL domains, including fatigue and depression. HU adherence will be measured using electronic pill bottles, self-report measures, laboratory markers, and medication possession ratio (MPR). HRQOL will be assessed using PROMIS® measures.

Hypothesis 2: Low HU adherence is associated with impairment of HRQoL domains.

Aim 3: Conduct a single-arm, pilot study to determine the effect size associated with improvement in HU adherence after using HU-Go for 12 weeks. Adherence will be measured using self-report measures, laboratory markers and MPR.

Hypothesis 3: HU-Go will improve HU adherence by at least 20%.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years old at the time of study enrollment
* Diagnosis of sickle cell disease (hemoglobin SS or SC or S/B 0 thalassemia) confirmed by hemoglobin electrophoresis
* On hydroxyurea
* Own or have access to a smartphone
* Be able to speak and read English

Exclusion Criteria:

* Chronic monthly transfusion support
* Any hemoglobinopathy other than sickle cell disease

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-11 (Actual)

PRIMARY OUTCOMES:
Achieving feasibility based on the number of participants completed all study procedures within 6 months of study enrollment | 3 months of study enrollment
  Feasibility is defined as having 80% or more of study participants complete the study within 6 months of enrollment

SECONDARY OUTCOMES:
Adherence to Hydroxyurea using Modified Morisky Adherence Scale 8-items | 3 months of study enrollment
  Numerical value on a scale 0-8 (higher score indicating higher adherence to hydroxyurea)
Adherence to Hydroxyurea using Visual Analogue Scale | 3 months of study enrollment
  Numerical value on a scale 0-100% (higher score indicating higher adherence to hydroxyurea)
Patient satisfaction with the smartphone app intervention (HU-Go) | 3 months of study enrollment
  Customized patient satisfaction questionnaire, numerical value on a scale 0-10 (higher score indicating higher satisfaction with the app)
HRQOL outcomes | 3 months
  Patient reported outcomes measurement information system (PROMIS) measures, numerical value on a scale of 0-100 points, normal average for the general population is 50 with standard deviation of 10 points. Each HRQOL outcome domain score will be reported separately (higher T scores indicating worse pain, fatigue, depression and anxiety, and lower scores indicating worse physical functioning and peer relationships).

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M. Badawy, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
All patients data will be deidentified.